CLINICAL TRIAL: NCT02443961
Title: Clinical Trial: Security and Feasibility of Mesenchymal Stem Cell Therapy in Treatment and Prevention of Bronchopulmonary Dysplasia in Preterm Babies
Brief Title: Mesenchymal Stem Cell Therapy for Bronchopulmonary Dysplasia in Preterm Babies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Fundación de Ayuda a la Investigación sobre la Hipertensión pulmonar (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PULMESCEL-1
Record Dates: First submitted 2015-05-04; First posted 2015-05-14 (Estimated); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary dysplasia; pulmonary hypertension; stem cell therapy; mesenchymal stem cells; very low weight preterm babies
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Hypertension, Pulmonary | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mesenchymal Stem Cell (MSC) therapy (Experimental): There will only be one treatment arm to evaluate the security of the treatment with MSC.
  Interventions: Biological: Mesenchymal Stem Cell (MSC) therapy

INTERVENTIONS:
Biological: Mesenchymal Stem Cell (MSC) therapy — 3 doses of 5 million MSC will be administered

SUMMARY:
Bronchopulmonary Dysplasia (BPD) is the most frequent disease related to a premature birth, 15-50% of very low birth newborns (<1500 gr.) will develop BPD. The prevalence of BPD is increasing due to the advances in neonatology, with a rise in the survival of smaller and more premature babies. The etiology of BPD is multifactorial, in which oxygen, maternal chorioamnionitis, insufficient pulmonary maturation etc. have an important role. These factors lead to a pathological development of the lung and pulmonary vessels, developing secondary Pulmonary Hypertension (PH). Nowadays there is no efficient treatment; this generates a important sanitary burden and a decrease in life quality. Multiple experimental models in mice have studied Mesenchymal Stem Cell (MSC) therapy as prevention of BPD, also recently some clinical trials have tried this therapy on premature newborns with promising results. Hypothesis: MSC therapy in patients at high risk of BPD prevents pulmonary lesions. Methods: The investigators have designed a clinical trial to evaluate the feasibility and security of MSC therapy in patients at high risk of developing BPD.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns ≤ 28 weeks gestational age
* Birth Weight <1250 gr.
* Still on of mechanical ventilation FiO2 > 0,3 at day + 14

Exclusion Criteria:

* Other congenital pathology (pulmonary malformations, active pulmonary bleeding, renal malformations, CHD, malformative syndromes, chromosomopathies)
* Severe neurological lesion.
* HIV infection
* Cardiovascular instability due to any cause
* 72 hours after mayor surgery
* Necrotizing enterocolitis grades II or higher, according to Bell classification, at the time of inclusion.

Ages: 1 Week to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-04-02 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and security of MSC therapy in very low birth weight preterm babies at risk of developing bronchopulmonary dysplasia (Number of participants with adverse events) | 24 months
  Number of participants with adverse events as a measure of safety and tolerability

SECONDARY OUTCOMES:
Biomarker analysis (IL-1beta, IL-6, IP-10, INF-gamma, TGF beta, NLRP3, RAGE, HMGB1, VEGFA, GREMLIN1, sVEGFR1, IGF, ENDOTHELIN-1, SMPD-1, SP-D, SMPD3. | 24 months
  biomarkers will be measured in pg/ml
Changes in the echocardiographic parameters related with PH and preterm birth, in patients treated with MSC (Number of participants with echocardiographic adverse events) | 24 months
  Flattening of the interventricular septum will be the main parameter (tipe I, I-II, II, II-III OR III)
Incidence of BPD and PH in very low birth weight babies treated with MSC | 24 months
  Diagnosed at 36 weeks of postmenstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jesus del Cerro, PhD, Principal Investigator — IRYCIS. Hospital Universitario Ramón y Cajal. Madrid. Spain
Locations (4):
- Spain (4):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No